CLINICAL TRIAL: NCT00633633
Title: Take Heart: Exercise & Diet Intervention for Heart Failure in Cancer Survivors
Brief Title: Lifestyle Intervention for Heart Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-0822; NCI-2011-02123 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Lifestyle Intervention; Exercise; Diet
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Usual Care
  Interventions: Other: Usual Care
- Group 2 (Experimental): Exercise Training + Dietary Counseling
  Interventions: Other: Usual Care; Behavioral: Exercise Training; Behavioral: Dietary Counseling

INTERVENTIONS:
Other: Usual Care — Monthly visits with the cardiology team and a booklet about coping with heart failure.
Behavioral: Exercise Training — Exercise training 3 times a week.
  Arms: Group 2
Behavioral: Dietary Counseling — Food log, booklet, and a cookbook to help decrease the salt content in your diet.
  Arms: Group 2

SUMMARY:
The goal of this behavioral research study is to learn if education and training about exercise can help to change the lifestyle of cancer survivors with symptoms of heart failure.

DETAILED DESCRIPTION:
Baseline Study Procedures:

If you agree to take part in the pretest portion of this study, your cardiology team will look at a number of tests performed on your heart as part of your usual care, as well as your complete medical history, to find out if you are eligible to take part in this study.

If you are found to be eligible to take part in this study, you will be scheduled for a visit to the Behavioral Research and Treatment Center (BRTC) at MD Anderson.

Before your first visit to the BRTC, you will complete the following tasks at home:

-You will wear an accelerometer to measure your physical activity for 1 week. An accelerometer is a small device that you wear on your waist during the day. It records how active you are. You will bring the accelerometer with you when you come for your first visit in the BRTC.

During your first visit to the BRTC, the following tests and procedures will be performed:

* You will have an electrocardiogram (ECG), which takes about 10 minutes. An ECG is a test used to measure the electrical activity of the heart.
* You will have your blood pressure and heart rate measured.
* You will complete questionnaires about your symptoms, quality-of-life, psychological distress, and exercise. These should take about 60 minutes to complete.
* You will complete 2 reaction time tasks on the computer. In one task, you will press a button on the keyboard to indicate the color of a word on the screen. In the other task, the computer will present a statement and you will press a button on the keyboard to indicate whether you think it is true or false. The statements are all opinions. It is not a test of knowledge. The 2 reaction time tasks together should take a total of about 10 minutes.
* You will do an exercise test on the stationary bicycle. You will ride on the stationary bicycle for about 10-15 minutes while your heart rate, blood pressure, and breathing are recorded by certified exercise specialists. While you are pedaling, the difficulty level will be changed by the study staff. First, you will pedal at a low difficulty level. After a 5-minute warm up period, the difficulty level will be slowly increased for about 3-5 minutes until you reach the point you cannot continue at that difficulty level. After that point, the difficulty level will be lowered for about 5 minutes to allow you to cool down. You can stop the test at any time.
* Then, you will repeat completing the exercise questionnaires and the reaction time tasks on the computer, which should take about another 10 minutes.

Study Groups:

After the above test and procedures, you will be randomly assigned (as in the flip of a coin) to be in 1 of 2 groups. You will have an equal chance of being in either group.

If you are in Group 1, you will receive the usual care as provided by the cardiology service, and a booklet about coping with heart failure. Dietary counseling will be provided once a month to encourage you to follow to a low sodium diet, with the goal of limiting sodium to 2 grams per day. The dietary counseling will include education about the effects of sodium for patients with heart failure, sources of sodium in the diet, reading food labels, identifying low-sodium alternatives to high-sodium foods, and using other types of flavorings rather than salt and other high-sodium condiments. You will be given the booklet How to Follow a Low Sodium Diet from the Heart Failure Society of America (appendix S and a copy of the American Heart Association Low-Salt Cookbook, 3rd edition. If you are a tobacco user or have recently quit, you will be referred to the MD Anderson Tobacco Treatment program. At the end of 16 weeks, after you have completed your 4 month visit in the BRTC, you will be offered exercise training described below. If you want to participate in the exercise training, you may do so at that time.

If you are in Group 2, you will receive all the components of usual care, plus exercise training.

Exercise Training:

If you are in Group 2, you will visit the BRTC 3 times a week for exercise training. For the first 12 sessions, you will exercise on a stationary bicycle while your heart rate, ECG, and blood pressure are recorded.

After the cardiologist finds that you are able to exercise safely, you will use part of the exercise session to do exercise without having your heart rate, ECG, and blood pressure recorded. Your exercise sessions at the BRTC will be supervised by a study staff member at all times. After you have exercised safely for at least 4 weeks, you will begin at-home exercise program, which will be a series of exercises developed individually for you, in addition to the supervised exercise sessions in the BRTC. You will be given an exercise log to describe your at-home exercise, and any problems or symptoms you experience during or after the at-home exercise sessions.

The visits to the BRTC for exercise training will last about 1 hour. You will come to the BRTC for these visits 3 times a week for 16 weeks.

If you are in Group 1, you have the option of choosing the exercise training described above or a 12-week home-based exercise training program that you will start after your 4 - month visit to the BRTC. You will be scheduled for an in-person exercise session with the exercise physiologist at the BRTC at MD Anderson. During this visit, you will receive instructions on how to complete your exercise sessions safely and effectively at home. This visit will take about 1 hour to complete. You will be provided with an exercise recommendation that will help you work up to 30 minutes of exercise, at least 3 times a week.

The exercise physiologist will call you once a week for 12 weeks to check on your progress and answer any questions you may have about your exercise program. You will also have the opportunity to come back to MD Anderson up to 1 time a week if you would like help from the exercise physiologist.

You will be given a pedometer to wear. A pedometer is a small device (about the size of a deck of cards) that is worn on the belt and measures the number of steps you take each day. You will record the number of steps and minutes of exercise for each day on an exercise log sheet.

At Weeks 4 and 8 (+/- 7 days), you will have a telephone interview about any side effects you may be having and how well you are able to function in daily activities.

You will also be counseled on limiting how much sodium you consume. The dietary counseling will include education about the effects of sodium on patients with heart failure, sources of sodium in the diet, reading food labels, identifying low-sodium alternatives to high-sodium foods, and using other types of flavorings rather than salt and other high-sodium condiments.

These calls should take about 45 minutes.

Follow-Up Visits:

If you are in either Group 1 or Group 2, you will have an appointment with the MD Anderson cardiology team 4 months from the baseline assessment. At this visit you will be asked about your symptoms. Blood (about 1 teaspoon) will be drawn to measure biomarkers at baseline and at the 4 month visit. Biomarkers are chemical "markers" in the blood that may be related to your heart failure.

If you are in Group 1 or Group 2, you will have a follow-up visit in the BRTC about 16-18 weeks after your baseline visit.

Ten (10) days before this visit, you will receive a new accelerometer in the mail. You will be called and reminded to wear the accelerometer. You will wear the accelerometer for 7 days and then bring it to the last visit to the BRTC.

At your last follow up visit to the BRTC, the following tests and procedures will be performed:

* You will complete questionnaires about your symptoms, quality of life, psychological distress, and exercise.
* You will complete 2 reaction time tasks on the computer.
* After these questionnaires and reaction tests, you will have an ECG and your blood pressure and heart rate will be measured.
* You will have an echocardiogram.
* You will then do an exercise test on the stationary bicycle.
* Then you will repeat the exercise questionnaires and the reaction time tasks on the computer.
* You will also be asked to take part in an interview about what you thought of the exercise program and the tasks you performed at home. This interview should take about 15 minutes.

After your 16-week visit, information about your cardiac tests, health problems, and hospitalizations will be collected from your medical record.

Participants in the waiting list group who choose to participate in the exercise program after their 16 week assessment will complete questionnaires once a month to measure symptoms. After 4 months of exercise (3 months for home-based) they will repeat all the follow-up tests described above.

This is an investigational study.

Up to 80 participants will be take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of NYHA I, II or III heart failure (as identified by any of the following physical findings of heart failure (jugular venous distension, crackles, edema, S3); pulmonary edema on chest x-ray; BNP > 100 pg/ml; or at least two of the following symptoms: paroxysmal nocturnal dyspnea, shortness of breath, swelling, fatigue;
2. previous chemotherapy that contributed to the development of heart failure (i.e., heart failure develops or worsens after receiving chemotherapy, with no other obvious explanation);
3. oriented to person, place, and time;
4. living in the Houston area (Harris county or a contiguous county), or planning to stay in the area for at least the next 16 weeks.
5. 18 years of age or older.
6. diagnosis of cancer
7. have completed treatment, or are on long-term adjuvant or maintenance chemotherapy only

Exclusion Criteria:

1. remain in NYHA class IV heart failure despite therapy;
2. have health problems or current treatments that would make exercise unsafe, as determined by the cardiologist;
3. cannot provide informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2008-02-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment/Attendance/Drop-Out Rates | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Tsai E, Mouhayar E, Lenihan D, Song J, Durand JB, Fadol A, Massey M, Harrison C, Basen-Engquist K. Feasibility and Outcomes of an Exercise Intervention for Chemotherapy-Induced Heart Failure. J Cardiopulm Rehabil Prev. 2019 May;39(3):199-203. doi: 10.1097/HCR.0000000000000388. PMID 31022003
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org